CLINICAL TRIAL: NCT04666038
Title: A Phase 3 Open-Label, Randomized Study of LOXO-305 Versus Investigator's Choice of Idelalisib Plus Rituximab or Bendamustine Plus Rituximab in BTK Inhibitor Pretreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (BRUIN CLL-321)
Brief Title: Study of LOXO-305 (Pirtobrutinib) Versus Investigator's Choice (Idelalisib Plus Rituximab or Bendamustine Plus Rituximab) in Patients With Previously Treated Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Acronym: BRUIN CLL-321
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18073; J2N-OX-JZNN (Other: Eli Lilly and Company); LOXO-BTK-20020 (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Hematologic Disease; Lymphoma, non-Hodgkin's; Lymphoma, B-cell; Lymphoma; Bruton's tyrosine kinase inhibitor; Ibrutinib; Acalabrutinib; Zanubrutinib; Pirtobrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Diseases; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma | interventions — pirtobrutinib; idelalisib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized in 1:1 into Arm A or Arm B. Patients randomized to Arm B who have disease progression (PD) confirmed by independent review committee (IRC) may be eligible to crossover into Arm A. Patients who discontinue treatment for toxicity may still be evaluated for cross over at the time of IRC-confirmed PD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Pirtobrutinib (Experimental): Participants received 200 milligrams (mg) of pirtobrutinib administered orally once daily (QD) on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
  Interventions: Drug: Pirtobrutinib
- Arm B - Idelalisib plus Rituximab or Bendamustine plus Rituximab (Active Comparator): Participants received either 150 mg of idelalisib administered twice-daily (BID) orally on Days 1 through 28 of a 28-day cycle in combination with 375 milligram per square meter (mg/m^2) of rituximab by intravenous (IV) infusion on day 1 of cycle 1, then 4 IV infusions of rituximab 500 mg/m^2 every 2 weeks (Q2W) and 3 IV infusions of rituximab 500 mg/m^2 every 4 weeks (Q4W) or 70 mg/m^2 of bendamustine administered IV on day 1 and 2 of each 28-day cycle from cycles 1 to 6 in combination with 375 mg/m^2 of rituximab IV on day 1 of cycle 1, then 500 mg/m^2 of rituximab on day 1 of each 28-day cycle from cycles 2 to 6.
  Interventions: Drug: Idelalisib; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Pirtobrutinib — Oral Pirtobrutinib
  Other Names: LOXO-305; LY3527727
  Arms: Arm A - Pirtobrutinib
Drug: Idelalisib — Oral
  Other Names: Zydelig
  Arms: Arm B - Idelalisib plus Rituximab or Bendamustine plus Rituximab
Drug: Bendamustine — IV
  Other Names: Treanda, Treakisym, Ribomustin, Levact
  Arms: Arm B - Idelalisib plus Rituximab or Bendamustine plus Rituximab
Drug: Rituximab — IV
  Other Names: Rituxan, MabThera, Truxima
  Arms: Arm B - Idelalisib plus Rituximab or Bendamustine plus Rituximab

SUMMARY:
This is a study for patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) who have previously received treatment with at least a BTK inhibitor. The main purpose is to compare LOXO-305 to idelalisib plus rituximab or bendamustine plus rituximab. Participation could last up to four years, and possibly longer, if the disease does not progress.

DETAILED DESCRIPTION:
This is a Phase 3 global, randomized, open-label study comparing LOXO-305 (Arm A) to investigator's choice of either idelalisib plus rituximab or bendamustine plus rituximab (Arm B) in CLL/SLL patients who have been treated with at least a covalent BTK inhibitor (BTKi). Patients may have discontinued the prior covalent BTKi due to disease progression (PD) or intolerance. Patients who have received venetoclax are eligible for the study. Eligible patients will be randomized in 1:1 to Arm A or Arm B.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL/SLL requiring therapy as defined by iwCLL 2018 criteria.
* Previously treated with a covalent BTK inhibitor.
* Eastern Cooperative Oncology Group (ECOG) 0-2.
* Absolute neutrophil count ≥ 0.75 × 10^9/L without granulocyte-colony-stimulating factor support, or ≥ 0.50 × 10^9/L in patients with documented bone marrow involvement considered to impair hematopoiesis. Granulocyte-colony-stimulating factor support is permitted in patients with documented bone marrow involvement.
* Hemoglobin ≥ 8 g/dL or ≥ 6 g/dL in patients with documented bone marrow involvement considered to impair hematopoiesis. Transfusion support is permitted in patients with bone marrow involvement.
* Platelets ≥ 50 × 10^9/L. If an investigator has chosen bendamustine/rituximab as the Arm B treatment, platelets must be ≥ 75 × 10^9/L. Patients may enroll below these thresholds if the Investigator determines the cytopenia is related to bone marrow involvement considered to impair hematopoiesis. Patients with a platelet count < 30 x 10^9/L are excluded.
* AST and ALT ≤ 3.0 x upper limit of normal (ULN).
* Total bilirubin ≤ 1.5 x ULN.
* Estimated creatinine clearance of ≥ 30 mL/min.

Exclusion Criteria:

* Known or suspected Richter's transformation at any time preceding enrollment.
* Known or suspected history of central nervous system (CNS) involvement by CLL/SLL.
* Ongoing drug-induced liver injury.
* Active uncontrolled auto-immune cytopenia.
* Significant cardiovascular disease.
* History of allogeneic or stem cell transplantation (SCT) or chimeric antigen receptor-modified T cells (CAR-T) therapy within the past 60 days.
* Active hepatitis B or hepatitis C.
* Known active cytomegalovirus (CMV) infection.
* Active uncontrolled systemic bacterial, viral, fungal or parasitic infection.
* Known Human Immunodeficiency Virus (HIV) infection, regardless of CD4 count.
* Clinically significant active malabsorption syndrome or inflammatory bowel disease
* Prior exposure to non-covalent (reversible) BTK inhibitor.
* Patients requiring therapeutic anticoagulation with warfarin or another Vitamin K antagonist.
* Current treatment with strong cytochrome P450 (CYP) 3A4 (CYP3A4) inhibitors or inducers.
* Vaccination with a live vaccine within 28 days prior to randomization.
* Patients with the following hypersensitivity:

  1. Known hypersensitivity, including anaphylaxis, to any component or excipient of LOXO-305. For patients planned to receive idelalisib, known hypersensitivity, including anaphylaxis, to any component or excipient of idelalisib. For patients planned to receive bendamustine, known hypersensitivity, including anaphylaxis, to any component or excipient of bendamustine.
  2. Prior significant hypersensitivity to rituximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2027-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Hill, MD, Study Director — Loxo Oncology, Inc.
Locations (232):
- United States (46):
  - Southern Cancer Center, P.C., Daphne, Alabama
  - Mitchell Cancer Institute -University of South Alabama, Mobile, Alabama
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Arizona Oncology Associates, P.C. - HOPE, Tucson, Arizona
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - California Research Institute, Los Angeles, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Cancer Specialists of North Florida -St Augustine, Jacksonville, Florida
  - Oncology-Hematology Associates of West Broward, Tamarac, Florida
  - WellStar Health System, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Arnett Cancer Center, Lafayette, Indiana
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Mercy Health-Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Cancer Center Office of Clinical Research, New Orleans, Louisiana
  - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Ascension St. John Hospital, Grosse Pointe Woods, Michigan
  - Minnesota Oncology/Hematology PA, Saint Paul, Minnesota
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Nebraska Hematology-Oncology, Lincoln, Nebraska
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Clinical Research Alliance, Inc., Westbury, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Oncology Fort Worth, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Roanoke, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Australia (7):
  - Canberra Hospital, Garran, Australian Capital Territory
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - The St. George Hospital, Kogarah, New South Wales
  - Ingham Institute of Medical Research, Liverpool, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - Uniklinikum Salzburg, Salzburg, Osterreich
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna
- Belgium (7):
  - CHR Verviers-Onco, Verviers, Liege
  - VITAZ, Sint-Niklaas, Oost-Vlaanderen
  - AZ Delta, Roeselare, West Flanders
  - Universitair Ziekenhuis Gent, Ghent
  - Groupe Jolimont, Haine-Saint-Paul
  - AZ St-Elisabeth, Herentals
  - Clinique Saint Pierre Ottignies, Ottignies
- Canada (4):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Princess Margaret Hospital (Ontario), Toronto, Ontario
- China (20):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Xicheng District, Beijing Municipality
  - Gansu Province Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Hainan Province People's Hospital, Haikou, Hainan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Taizhou Hospital, Linhai, Zhejiang
  - Beijing Hospital, Beijing
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Blood Institute of the Chinese Academy of Medical science, Tianjin
- Croatia (2):
  - University Hospital Split, Split
  - Division of Hematology, Dept. of Internal Medicine, University Hospital Centre Zagreb, Zagreb
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (14):
  - CHU De Grenoble Hopital Albert Michallon, Grenoble, Cedex 09
  - Hospital AVICENNE, Bobigny, Cedex
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Cedex
  - CHD Vendee, La Roche-sur-Yon, La Roche Sur Yon
  - Chu Nimes/Institut De Cancerologie Du Gard, Nîmes, Nimes
  - Pole Regionalde Cancérologie(CHU de Poitiers), Politiers, Politiers
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen, Rouen, Seine-Maritime
  - CHRU De Tours, Tours, Tours Cedex 9
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - CHRU de Brest - Hôpital Morvan, Brest
  - Centre Hospitalier du Mans, Le Mans
  - Hopital Saint Vincent De Paul, Lille
  - Ch Perpignan, Perpignan
- Germany (8):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Uniklinik Köln, Kerpener, Köln
  - Universitätsmedizin Mainz III. Medizinische Klinik und Poliklinik, Langenbeckstraße 1, Mainz
  - München Klinik Schwabing, Koelner Platz 1, München
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Lübecker Onkologische Schwerpunktpraxis, Lübeck, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum, Berlin
- Hungary (4):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - University of Pecs 1st. Internalmedicin Clinic Dept, Pécs
- Ireland (3):
  - St James's Hosptial, Dublin
  - Beaumont Hospital, Dublin, Dublin
  - Mater Misericordiae Hospital, Dublin
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - Soroka Medical Center, Beersheba
  - Laniado Medical Center, Netanya
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Carmel Hospital, Haifa, Ḥeifā
- Italy (25):
  - Irccs Istituto Tumori Giovanni Paolo Ii, Viale Orazio Flacco, Bari
  - ASST-Monza -U.O Ematologia Adulti, Monza (MB) -Settore E, Piano 2
  - Azienda Ospedaliero Universitaria Pisana, Pisa, PI
  - Irccs Crob, Rionero in Vulture, Potenza
  - AULSS8 Berica-Ospedale S.Bortolo, Vicenza, Veneto
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - ASST Spedali Civili - Università degli Studi, Brescia
  - A.O.U. Policlinico G.Rodolico - S. Marco, Catania
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Papardo, Messina
  - IRCCS Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda Comitato Etico Milano Area C, Milan
  - A.O.U. di Modena, Modena
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Istituto di Ematologia-C.R.E.O. (Centro di Ricerche Emato-Oncologich), Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Santa Maria Terni, Terni
  - A.O.U. Citta' della Salute e della Scienza di Torino, Torino
  - Az. Osp. "Card G Panico", Tricase
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
  - Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona
- Japan (18):
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tokai University Hospital- Isehara Campus, Isehara, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Tohoku University Hospital, Sendai, Miyagi
  - NHO Sendai Medical Center, Sendai, Miyagi
  - Kindai University Hospital, Osaka Sayama-shi, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-Ku, Tokyo
  - JCHO Kyushu Hospital, Fukoka-ken
  - Kumamoto University Hospital, Kumamoto
  - Okayama University Hospital, Okayama
  - Osaka University Hospital, Osaka
- Poland (13):
  - Wojewodzki Szpital Specjalistyczny, Iwaszkiewicza 5, Legnica
  - Centrum Onkologii Ziemi Lubelskiej, Lublin, Lublin Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Szpitale Pomorskie Sp. z o. o., Gdynia, Pomeranian Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny im.ks.B.Markiewicza, Brzozów
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w BydgoszczyKlinika Hematologii, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii, Lodz
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
  - Oddzial Hematologiczny, Specjalistyczny Szpital im. dra Sokołowskiego w Wałbrzychu, Wałbrzych
  - Uniwersytecki Szpital Kliniczny Klinika, Wroclaw
- Russia (4):
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncology Dispensary", Omsk, Omsk Oblast
  - Federal State Budgetary Institution "Russian Scientific and Research Institute of Hematology and Transfusiology of Federal Medico-Biological Agency, Saint Petersburg
  - Academician I.P. Pavlov First St-Petersburg State Medical University, Saint Petersburg
  - Oncology Dispensary #2 of Krasnodar Region, Sochi
- Gleneagles Medical Centre, Singapore, Central Singapore, Singapore
- South Korea (6):
  - Gachon University Gil Hospital, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - Pusan National University Hospital, Busan, Pusan-Kwangyǒkshi
  - The Catholic University of Korea-Seoul St. Mary's Hospital, Seocho-Gu, Seoul
  - Seoul National University Hospital, Seoul, Seoul, Korea
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Inje Univ Busan Paik Hospital, Busan
- Spain (15):
  - Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Toledo, Toledo, Castille-La Mancha
  - Complejo Hospitalario Universitario de Santiago de Compostel, Santiago de Compostela, La Coruna
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid, Comunidad de
  - Hospital General Universitario Gregorio Marañón, Madrid, Planta Baja
  - Hospital General de Albacete, Albacete
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Infanta Leonor-INTERNAL MED, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Marques De Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario de Alava, Vitoria-Gasteiz
- Clinica di Ematologia IOSI, Ospedale Bellinzona e Valli, Ente Ospedaliero Cantonale, Bellinzona, Svizzera, Switzerland
- Taiwan (4):
  - China Medical University Hospital, Taichung, Taichung
  - Tri-Service General Hospital, Taipei City, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan, (r.o.c.), Taiwan
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Ankara University Medicine Hospital, Mamak, Ankara
  - Istanbul University Istanbul Medicine Faculty, Faith, Istanbul
  - Erciyes University Faculty of Medicine, Kayseri, Melikgazi
  - Gazi University Faculty of Medicine, Ankara, Yenimahalle
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Faculty of Medicine, Izmir
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeen City
  - The Royal Cornwall Hospital, Truro, Cornwall
  - Derriford Hospital, Plymouth, Devon
  - Castle Hill Hospital, Cottingham, East Yorkshire
  - University College London Hospitals, London, Greater London
  - Norfolk and Norwich Hospital, Norwich, Norfolk
  - Singleton Hospital, Swansea, SA2 8QA
  - Western General Hospital, Edinburgh, Scotland
  - Royal Marsden Hospital, Sutton, Surrey
  - St Johns Hospital at Howden, Livingston, West Lothian
  - St James's University Hospital, Leeds
  - Milton Keynes University Hospital, Milton Keynes
  - GenesisCare Cambridge, Newmarket

REFERENCES:
- [Derived] Sharman JP, Munir T, Grosicki S, Roeker LE, Burke JM, Chen CI, Grzasko N, Follows G, Matrai Z, Sanna A, Qiu L, Feng R, Hua VM, Jurczak W, Ritgen M, Yi S, Bosch F, Coombs CC, Bao K, Patel V, Liu B, Compte L, Guntur A, Wang DY, Hill M, Leow CC, Ghia P, Barr PM. Phase III Trial of Pirtobrutinib Versus Idelalisib/Rituximab or Bendamustine/Rituximab in Covalent Bruton Tyrosine Kinase Inhibitor-Pretreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (BRUIN CLL-321). J Clin Oncol. 2025 Aug;43(22):2538-2549. doi: 10.1200/JCO-25-00166. Epub 2025 Jun 6. PMID 40479620

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 238 participants were randomized 1:1 to receive either Arm A - pirtobrutinib or Arm B - Idelalisib plus Rituximab or Bendamustine plus Rituximab. The results were reported based on a data cut off from 29 Aug 2024.
Period: Overall Study
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Started | 119 | 119
Received at Least 1 Dose of Study Drug | 116 | 109
Completed | 0 | 0
Not Completed | 119 | 119
Not completed — Progressive Disease | 2 | 0
Not completed — Death | 38 | 32
Not completed — Withdrawal by Subject | 10 | 19
Not completed — Lost to Follow-up | 0 | 2
Not completed — On Study Treatment | 46 | 5
Not completed — Off treatment on post-treatment-discontinuation follow-up | 23 | 61

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Arm A - Pirtobrutinib: Participants received 200 mg of pirtobrutinib administered orally QD on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
- Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab: Participants received either 150 mg of idelalisib administered BID orally on Days 1 through 28 of a 28-day cycle in combination with 375 mg/m^2 of rituximab by IV infusion on day 1 of cycle 1, then 4 IV infusions of rituximab 500 mg/m^2 Q2W and 3 IV infusions of rituximab 500 mg/m^2 Q4W or 70 mg/m^2 of bendamustine administered IV on day 1 and 2 of each 28-day cycle from cycles 1 to 6 in combination with 375 mg/m^2 of rituximab IV on day 1 of cycle 1, then 500 mg/m^2 of rituximab on day 1 of each 28-day cycle from cycles 2 to 6.
- Total: Total of all reporting groups
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab | Total
Number analyzed (Participants) | 119 | 119 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.90 (9.32) | 67.00 (8.52) | 67.00 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 83 | 83 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 107 | 108 | 215
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 98 | 95 | 193
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 2 | 7
  Austria | 1 | 1 | 2
  Belgium | 1 | 0 | 1
  Canada | 4 | 6 | 10
  China | 10 | 14 | 24
  Croatia | 0 | 1 | 1
  Czechia | 2 | 1 | 3
  France | 5 | 4 | 9
  Germany | 2 | 4 | 6
  Hungary | 3 | 4 | 7
  Ireland | 2 | 1 | 3
  Israel | 2 | 0 | 2
  Italy | 23 | 19 | 42
  Japan | 3 | 0 | 3
  Poland | 14 | 17 | 31
  Russia | 0 | 1 | 1
  South Korea | 1 | 0 | 1
  Spain | 4 | 2 | 6
  Switzerland | 2 | 1 | 3
  Taiwan | 0 | 1 | 1
  Turkey | 1 | 1 | 2
  United Kingdom | 14 | 6 | 20
  United States | 20 | 33 | 53

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Assessed by Independent Review Committee (IRC)
Description: PFS is defined as the time from the date of randomization to the date of first documentation of progressive disease (PD) or death from any cause, as evaluated by an IRC according to International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018.
Time Frame: Randomization to Disease Progression or Death Due to Any Cause (Up to 29 Months)
Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 119 | 119
Months | 13.96 [11.24 to 16.56] | 8.74 [8.08 to 10.38]
Statistical Analysis 1: Comparison: Arm A - Pirtobrutinib vs Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab; Test type: Superiority; p = 0.0002, Log Rank — The 2-sided nominal p-value was calculated based on a stratified log-rank test; Hazard Ratio (HR) = 0.536, 95% CI 2-sided [0.385 to 0.746] — The Hazard Ratio (HR) & 95% confidence interval (CI) were estimated from a stratified Cox proportional hazards model

2. Secondary Outcome: PFS Assessed by Investigator
Description: PFS is defined as time from the date of randomization to the date of first documentation of PD or death from any cause, as evaluated by an investigator according to iwCLL 2018.
Time Frame: Randomization to Disease Progression or Death Due to Any Cause (Up to 36 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 119 | 119
Months | 15.28 [12.81 to 19.94] | 9.20 [7.33 to 10.64]
Statistical Analysis 1: Comparison: Arm A - Pirtobrutinib vs Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab; Test type: Superiority; p < 0.0001, Log Rank — The 2-sided nominal p-value was calculated based on a stratified log-rank test; Hazard Ratio (HR) = 0.475, 95% CI 2-sided [0.338 to 0.669] — The HR and 95% CI were estimated from a stratified Cox proportional hazards model

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from randomization to death due to any cause.
Time Frame: Randomization to Death from Any Cause (Up to 36 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 119 | 119
Months | 29.67 [27.10 to NA] — Median estimate is unstable due to few patients at risk at later time points. Upper limit of 95% CI was not estimable due to low number of participants with events (events = 38). | NA [28.88 to NA] — Median and upper limit of 95% CI was not estimable due to low number of participants with events (events = 32).
Statistical Analysis 1: Comparison: Arm A - Pirtobrutinib vs Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab; Test type: Superiority; p = 0.7202, Log Rank — The 2-sided p-value was calculated based on a stratified log-rank test; Hazard Ratio (HR) = 1.090, 95% CI 2-sided [0.679 to 1.749] — The HR and 95% CI were estimated from a stratified Cox proportional hazards model

4. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT was defined as time from the date of randomization to the date of initiation of the subsequent anticancer therapy for chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), therapy of pirtobrutinib for Arm B patients, or death due to any cause, whichever occurs first.
Time Frame: Randomization to Subsequent Anticancer Therapy, Therapy of Pirtobrutinib or Death Due to Any Cause (Up to 36 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 119 | 119
Months | 23.95 [17.84 to 29.67] | 10.91 [8.74 to 12.48]
Statistical Analysis 1: Comparison: Arm A - Pirtobrutinib vs Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab; Test type: Superiority; p < 0.0001, Log Rank — The 2-sided nominal p-value was calculated based on a stratified log-rank test; Hazard Ratio (HR) = 0.365, 95% CI 2-sided [0.254 to 0.524] — The HR and 95% CI were estimated from a stratified Cox proportional hazards model

5. Secondary Outcome: Event Free Survival (EFS)
Description: EFS is defined as the time from randomization to the first occurrence of:
  * Documented disease progression per iwCLL 2018 criteria as assessed by Investigator; or
  * Initiation of subsequent anticancer therapy for CLL/SLL; or
  * Unacceptable toxicity leading to treatment discontinuation as assessed by the Investigator; or
  * Death (due to any cause).
Time Frame: Randomization to Disease Progression, Subsequent Anticancer Therapy, Unacceptable Toxicity Leading to Treatment Discontinuation, or Death Due to Any Cause (Up to 36 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 119 | 119
Months | 14.06 [11.40 to 16.95] | 7.62 [4.80 to 8.80]
Statistical Analysis 1: Comparison: Arm A - Pirtobrutinib vs Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab; Test type: Superiority; p < 0.0001, Log Rank — The 2-sided nominal p-value was calculated based on a stratified log-rank test; Hazard Ratio (HR) = 0.387, 95% CI 2-sided [0.280 to 0.534] — The HR and 95% CI were estimated from a stratified Cox proportional hazards model

6. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR) Assessed by Investigator
Description: ORR according to investigator-assessed best overall response (BOR) based on iwCLL 2018 is defined as the number of participants who achieve a BOR of complete response (CR), complete response with incomplete bone marrow recovery (CRi), nodular partial response (nPR) or partial response (PR) at or before the initiation of subsequent anticancer therapy divided by the total number of participants randomized to each treatment arm.
Time Frame: Randomization to Subsequent Anticancer Therapy, Disease Progression or Death Due to Any Cause (Up to 36 Months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 119 | 119
percentage of participants | 66.4 [57.15 to 74.78] | 48.7 [39.47 to 58.07]

7. Secondary Outcome: Time to Worsening (TTW) of CLL/SLL Related Symptoms
Description: TTW was defined as a change in score greater than the meaningful within-person change for worsening in score. Scores were furthermore required to be sustained. To meet the requirement for sustained change, the assessment following the first observation of a meaningful worsening of the score (event date) was also required to show a meaningful worsening compared to baseline. The event date was defined as the first of these consecutive events. The European Organization for Research and Treatment of Cancer Item Library 87 was used, which is scored from 0-100, with higher scores reflecting more symptoms.
  The time to sustained patient-reported outcome (PRO) deterioration was calculated using all on-treatment assessment time points up to the Week 25 (Arm A & Arm B - Idelalisib plus Rituximab) and up to Week 21 + Safety follow-up of up to 5 weeks (Arm B - Bendamustine plus Rituximab) assessment time point prior to disease progression.
Time Frame: Baseline up to Week 25 (Arm A and Arm B - Idelalisib plus Rituximab) & Baseline up to Week 21 + Safety Follow-Up of up to 5 Weeks (Arm B - Bendamustine plus Rituximab)
Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 110 | 90
Months | NA [NA to NA] — Median and 95% CI was not estimable due to low number of events (events = 17). | NA [5.7 to NA] — Median and upper limit of 95% CI was not estimable due to low number of events (events = 11).

8. Secondary Outcome: Time to Worsening (TTW) of Physical Function
Description: Time of worsening was defined as a change in score greater than the meaningful within-person change for worsening in score. Scores were furthermore required to be sustained. To meet the requirement for sustained change, the assessment following the first observation of a meaningful worsening of the score (event date) was also required to show a meaningful worsening compared to baseline. The event date was defined as the first of these consecutive events. The European Organization for Research and Treatment of Cancer Item Library 87 was used, which is scored from 0-100, with higher scores reflecting more symptoms.
  The time to sustained PRO deterioration was calculated using all on-treatment assessment time points up to the Week 25 (Arm A and IdelaR) and up to Week 21 + Safety follow-up (BR) assessment time point prior to disease progression.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
Number analyzed (Participants) | 110 | 90
Months | NA [NA to NA] — Median and 95% CI was not estimable due to low number of events (events = 12). | NA [5.7 to NA] — Median and upper limit of 95% CI was not estimable due to low number of events (events = 11).

ADVERSE EVENTS:
Time Frame: Baseline up to data cut-off date 29-August-2024 (up to 36 months)
Description: All-Cause Mortality: All randomized participants. Serious and other adverse events: All randomized participants who received at least one dose of study drug; Analyses presented in this report were based on a data cut off from 29 Aug 2024. For Arm B, adverse events were presented for Investigator's choice of Idelalisib Plus Rituximab (IR) or Bendamustine Plus Rituximab (BR) combined. Arm B adverse event data was not collected separately for IR and BR.
Arm/Group | Arm A - Pirtobrutinib | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab
All-Cause Mortality (participants affected / at risk) | 38/119 | 32/119
Serious Adverse Events (participants affected / at risk) | 60/116 | 53/109
Other Adverse Events (participants affected / at risk) | 94/116 | 103/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A - Pirtobrutinib (N=116) | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab (N=109)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 2 (3)
Bone marrow necrosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (5)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 1 (2)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 6 (6)
Covid-19 pneumonia (Infections and infestations) | 5 (7) | 4 (4)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 20 (29) | 12 (15)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1/32 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/34 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Pirtobrutinib (N=116) | Arm B - Idelalisib Plus Rituximab or Bendamustine Plus Rituximab (N=109)
Anaemia (Blood and lymphatic system disorders) | 21 (29) | 21 (28)
Neutropenia (Blood and lymphatic system disorders) | 21 (44) | 17 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (13) | 7 (9)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 8 (10)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 8 (9)
Constipation (Gastrointestinal disorders) | 8 (9) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 20 (25) | 30 (45)
Nausea (Gastrointestinal disorders) | 13 (15) | 23 (37)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 8 (11)
Vomiting (Gastrointestinal disorders) | 7 (10) | 18 (26)
Asthenia (General disorders) | 10 (12) | 6 (10)
Chills (General disorders) | 1 (2) | 9 (9)
Fatigue (General disorders) | 16 (19) | 27 (29)
Oedema peripheral (General disorders) | 13 (15) | 7 (8)
Pyrexia (General disorders) | 14 (21) | 28 (35)
Bronchitis (Infections and infestations) | 3 (3) | 8 (11)
Covid-19 (Infections and infestations) | 14 (17) | 18 (21)
Pneumonia (Infections and infestations) | 15 (17) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 11 (18) | 7 (8)
Urinary tract infection (Infections and infestations) | 8 (13) | 4 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 16 (21)
Alanine aminotransferase increased (Investigations) | 4 (5) | 18 (29)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 13 (23)
Blood creatinine increased (Investigations) | 7 (8) | 8 (8)
Neutrophil count decreased (Investigations) | 9 (18) | 19 (41)
Platelet count decreased (Investigations) | 2 (6) | 13 (24)
Weight decreased (Investigations) | 4 (5) | 18 (19)
White blood cell count decreased (Investigations) | 2 (2) | 10 (34)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 15 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (10) | 4 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (10) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 5 (8)
Dizziness (Nervous system disorders) | 3 (3) | 9 (9)
Headache (Nervous system disorders) | 13 (14) | 15 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 20 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 11 (12) | 9 (11)
Hypertension (Vascular disorders) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT04666038/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04666038/SAP_001.pdf